CLINICAL TRIAL: NCT00630370
Title: A Phase II, Randomized, Adaptive Design, Multicenter, Parallel Group, Placebo-Controlled, 58 Day, Dose-Ranging Study of ATI 7505 in Patients With Postprandial Distress Syndrome
Brief Title: A Dose-Ranging Study of ATI 7505 in Patients With Postprandial Distress Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Collaborators: ARYx Therapeutics (Industry)
Responsible Party: Bruce Yacyshyn, MD, Procter & Gamble
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2007033
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2008-12

CONDITIONS: Post Prandial Distress Syndrome
MeSH Terms: interventions — ATI 7505

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): 2 Placebo tablets, TID, orally, 58 days
  Interventions: Drug: Placebo
- 2 (Experimental): 1 ATI 20mg and 1 placebo tablet, TID, orally, 58 days
  Interventions: Drug: 20 mg ATI 7505
- 3 (Experimental): 1 ATI 40mg and 1 placebo tablet, TID, orally, 58 days
  Interventions: Drug: 40 mg ATI 7505
- 4 (Experimental): 2 ATI 40mg tablets, TID, orally, 58 days
  Interventions: Drug: 80 mg ATI 7505

INTERVENTIONS:
Drug: Placebo — 2 Placebo tablets, TID, orally, 58 days
  Arms: 1
Drug: 20 mg ATI 7505 — 1 ATI 20mg and 1 placebo tablet, TID, orally, 58 days
  Arms: 2
Drug: 40 mg ATI 7505 — 1 ATI 40mg and 1 placebo tablet, TID, orally, 58 days
  Arms: 3
Drug: 80 mg ATI 7505 — 2 ATI 40mg tablets, TID, orally, 58 days
  Arms: 4

SUMMARY:
To assess the efficacy of 3 oral dosing regimens of ATI 7505 compared to placebo in patients with PDS by comparing at the end of Day 42 the percentage of patients in each treatment group who have had adequate relief of postprandial distress syndrome symptoms on at least 50% of the treatment days.

ELIGIBILITY:
Inclusion Criteria:

* Were diagnosed with PDS at least 6 months prior to screening, OR had onset of 2 or more PDS symptoms at least 6 months prior to screening.
* Experienced early satiety or bothersome postprandial fullness repeatedly during the 3 months prior to screening.
* Had a normal upper GI endoscopy within the past year.

Exclusion Criteria:

* Heartburn that occurs >3 times per week
* Current Helicobacter pylori (H pylori) infection confirmed by stool sample testing or breath testing, or H pylori eradication therapy within the 6 months prior to screening
* Any alarm symptoms including uninvestigated anemia, rectal bleeding, weight loss, or unresolved fever within the 6 months prior to screening
* At screening, a QT interval corrected for heart rate using Bazett's correction formula (QTcB) >440 msec as determined by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of 3 oral dosing regimens of ATI 7505 vs. placebo in patients with PDS. | Day 42

SECONDARY OUTCOMES:
Safety and tolerability of ATI 7505 | 42 days
Time to recurrence of the 2 primary PDS symptoms at day 42 | 42 days
Effect of ATI 7505 treatment on quality of life indices | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Bruce C Yacyshyn, MD, Study Director — Procter and Gamble
Locations (57):
- United States (40):
  - Research Facility, Chino, California
  - Research Facility, Fresno, California
  - Research Facility, Los Angeles, California
  - Research Facility, Mission Viejo, California
  - Research Facility, San Carlos, California
  - Research Facility, San Diego, California
  - Research Facility, Littleton, Colorado
  - Research Facility, Boynton Beach, Florida
  - Research Facility, DeLand, Florida
  - Research Facility, Hollywood, Florida
  - Research Facility, Jacksonville, Florida
  - Research Facility, Largo, Florida
  - Research Facility, Miami, Florida
  - Research Facility, New Port Richey, Florida
  - Research Facility, Orlando, Florida
  - Research Facility, Newnan, Georgia
  - Research Facility, Savannah, Georgia
  - Research Facility, Rockford, Illinois
  - Research Facility, Evansville, Indiana
  - Research Facility, Topeka, Kansas
  - Research Facility, Monroe, Louisiana
  - Research Facility, Detroit, Michigan
  - Research Facility, Brooklyn, New York
  - Research Facility, Great Neck, New York
  - Research Facility, Lake Success, New York
  - Research Facility, Syracuse, New York
  - Research Facility, Fayetteville, North Carolina
  - Research Facility, Winston-Salem, North Carolina
  - Research Facility, Cincinnati, Ohio
  - Research Facility, Dayton, Ohio
  - Research Facility, Oklahoma City, Oklahoma
  - Research Facility, Ashland, Oregon
  - Research Facility, Beaver Falls, Pennsylvania
  - Research Facility, Anderson, South Carolina
  - Research Facility, Charleston, South Carolina
  - Research Facility, Chattanooga, Tennessee
  - Research Facility, Colleyville, Texas
  - Research Facility, Salt Lake City, Utah
  - Research Facility, Winchester, Virginia
  - Research Facility, Milwaukee, Wisconsin
- Canada (9):
  - Research Facility, Guelph
  - Research Facility, Hamilton
  - Research Facility, Lévis
  - Research Facility, Longueuil
  - Research Facility, Montreal
  - Research Facility, Ottawa
  - Research Facility, Québec
  - Research Facility, Saint-Charles-Borromée
  - Research Facility, Toronto
- United Kingdom (8):
  - Research Facility, Birmingham
  - Research Facility, Cardiff
  - Research Facility, Coventry
  - Research Facility, Crewe
  - Research Facility, London
  - Research Facility, Norwich
  - Research Facility, Orpington
  - Research Facility, Salford